CLINICAL TRIAL: NCT00519974
Title: Decision-Making About Breast Reconstruction After Mastectomy Among Ethnic Minority Women: An Exploratory Study of Qualitative Themes
Brief Title: Factors Affecting Decisions About Breast Reconstruction After Mastectomy in Black and Latina Women
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07-087; P30CA008748 (NIH); MSKCC-07087
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: counseling intervention
Other: study of socioeconomic and demographic variables
Procedure: management of therapy complications
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Learning about the reasons for choosing to have, or not to have, breast reconstruction after mastectomy for breast cancer may help doctors understand why black or Latina women may or may not undergo breast reconstruction.

PURPOSE: This clinical trial is studying factors affecting decisions about breast reconstruction after mastectomy in black and Latina women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Interview black and Latina women about their reasons for choosing to have, or not to have, breast reconstruction after mastectomy for breast cancer.
* Describe the context in which black and Latina women make decisions about breast reconstruction.
* Explore similarities and differences in factors affecting decision-making among black and Latina women.
* Identify factors that contribute to the low utilization of breast reconstruction among ethnic minority women.

OUTLINE: This is a multicenter study.

Patients undergo a 1-hour interview to evaluate their rationale for choosing to have, or not to have, breast reconstruction after mastectomy. Interviews are conducted by a woman of the same ethnic background as the patient. Key factors influencing a patient's decision to consider having breast reconstruction are explored during the interview, including availability of educational materials on breast reconstruction and the adequacy of this information. Patients are asked to examine personal factors influencing their decision, such as feelings about living with or without a reconstructed breast; concerns about reconstructive surgery and its risks; potential complications; and impact of reconstructive surgery on sexuality and body image. Social and cultural factors are also evaluated, including influence of family and friends; degree of support for the patient's decision to have surgery; racial or ethnic differences in patient's preferences; and cultural values. Access-related factors, such as financial cost, insurance availability, or physician referral practices, are also explored.

At the end of the interview, patients may be referred to Memorial Sloan-Kettering Cancer Center or Ralph Lauren Center for Cancer Care and Prevention for oncologic surveillance or for additional information on breast reconstruction. Patients may also be contacted after the interview to answer follow-up questions, to clarify topics previously discussed, or to provide further input or feedback on preliminary study findings.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Have undergone mastectomy* (with or without reconstruction) for breast cancer within the past 3 years AND meets 1 of the following criteria:

  * Self-identified as being black
  * Self-identified as being Latina NOTE: *Patients scheduled to undergo mastectomy are eligible
* Recruited from one of the following cancer centers or breast cancer support organizations:

  * Memorial Sloan-Kettering Cancer Center or Ralph Lauren Center for Cancer Care and Prevention

    * Patients are identified by their physician (e.g., oncologist, breast surgeon), the protocol investigator, a member of the research team, and/or medical chart review
  * Spirit of Hope or LatinaSHARE

    * Patients are identified by the director of the support organization or the support group leader
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* No cognitive impairment that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Black and Latina female breast cancer patients who have undergone or scheduled to undergo mastectomy within the past 3 years will be identified by their physicians (e.g., medical oncologists, breast surgeon, plastic surgeon) at MSKCC and RLCCCP or by the advocacy center to which they belong.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Self-reported reasons among black and Latina women for choosing to have, or not to have, breast reconstruction after mastectomy | 2 years
Development of a theoretical model that describes how black and Latina women make decisions regarding breast reconstruction after mastectomy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L. Pusic, MD, MHS, Principal Investigator — Memorial Sloan Kettering Cancer Center; Karen Hurley, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - New School for Social Research, New York, New York
  - Spirit of Hope, New York, New York
  - Ralph Lauren Center for Cancer Care and Prevention, New York, New York
  - SHARE, Incorporated, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York